CLINICAL TRIAL: NCT06044077
Title: A Randomized, Blinded, Parallel Controlled Phase 3 Clinical Trial to Evaluate the Immunogenicity and Safety of the 23-valent Pneumococcal Polysaccharide Vaccine in Healthy People Aged 2 Years and Above
Brief Title: A Clinical Trial to Evaluate the Immunogenicity and Safety of the 23-valent Pneumococcal Polysaccharide Vaccine in Healthy People
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aimei Vacin BioPharm (Zhejiang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AM2022PPV23III
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 1 dose vaccination of study vaccine
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine
- Control Group (Other): 1 dose vaccination of control vaccine
  Interventions: Biological: control pneumococcal polysaccharide vaccine

INTERVENTIONS:
Biological: 23-valent pneumococcal polysaccharide vaccine — 23-valent pneumococcal polysaccharide vaccine from Aimei Vacin BioPharm (Zhejiang) Co., Ltd.
  Arms: Experimental Group
Biological: control pneumococcal polysaccharide vaccine — 23-valent pneumococcal polysaccharide vaccine from Merck Sharp & Dohme Corp
  Arms: Control Group

SUMMARY:
This study is a randomized, blinded, parallel controlled phase 3 clinical trial to evaluate the immunogenicity and safety of the 23-valent pneumococcal polysaccharide vaccine in healthy people aged 2 years and above.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects who meet the observation age of this clinical trial (2 years old and above) and are determined based on medical history, physical examination and the researcher's judgment;
2. Subjects who voluntarily participate and/or the subjects' legal guardians Or the entrusted person voluntarily agrees for his or her child to participate and signs an informed consent form (subjects aged 8-17 years old must also sign an informed notification form);
3. The subject and/or the subject's legal guardian or principal can abide by the clinical Relevant requirements of the research protocol;
4. *Axillary body temperature <37.3°C on the day of enrollment. For criteria marked with an asterisk (*), if the subject has the conditions specified in the criterion, the visit can be rescheduled when they no longer have those conditions.

Exclusion Criteria:

1. Previous vaccination with marketed or experimental pneumococcal vaccines;
2. Previous culture-confirmed history of invasive diseases caused by pneumococcal bacteria;
3. History or family history of convulsions, epilepsy, encephalopathy, and mental illness;
4. Have a history of severe allergy to any vaccination or drug in the past, be allergic to the ingredients of the experimental vaccine (mainly including pneumococcal polysaccharide, sodium dihydrogen phosphate, disodium hydrogen phosphate, and sodium chloride), and have a history of vaccination-related fever (39℃ or above );
5. Known severe congenital malformations, developmental disabilities or clinically diagnosed serious chronic diseases (such as Down syndrome, diabetes that cannot be controlled by drugs, sickle cell anemia, Guillain-Barré syndrome);
6. Known or suspected to have serious diseases including: severe respiratory diseases, severe digestive system diseases, severe endocrine system diseases, severe cardiovascular diseases, severe liver and kidney diseases, malignant tumors, severe skin diseases, etc.;
7. Known or suspected to be immune Academic functional defects include: immunosuppressant treatment (radiotherapy, chemotherapy, corticosteroids, antimetabolites, cytotoxic drugs), HIV infection, etc. within 6 months;
8. Have received any treatment within 3 months before enrollment Blood products or globulin treatment, those who have used hepatitis B immune globulin are acceptable;
9. Asplenia, functional asplenia or splenectomy;
10. * In the acute infectious period (including recovery period) or acute exacerbation of chronic disease within 3 days before enrollment, or need or plan to use intravenous or oral steroids within 1 month after vaccination;
11. * Antipyretic analgesics or anti-allergic drugs have been used within 3 days before enrollment;
12. Women of childbearing age are pregnant ( Positive urine pregnancy test), breastfeeding or planning to prepare for pregnancy within six months; 13. *Hypertension that cannot be controlled by medication, such as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg in adults aged 18 years and above before enrollment;

14. * Have received attenuated live vaccines within 14 days before vaccination, and received inactivated vaccines within 7 days; 15. Are participating in or plan to participate in clinical studies of other drugs or vaccines within 6 months after vaccination (immune persistence observation subjects in the vaccine who plan to vaccinate any marketed or unmarketed pneumococcal vaccine within 6 years after vaccination need to be excluded); 16. The investigators evaluate that they are not suitable for participating in the study.

For criteria marked with an asterisk (*), if the subject has the conditions specified in the criterion, the visit can be rescheduled when they no longer have those conditions.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1920 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-03-08 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
2-fold growth rate of IgG antibodies to 23 pneumococcal serotypes on 30 days after vaccination, | 30 days
  2-fold growth rate of IgG antibodies to 23 pneumococcal serotypes on 30 days after vaccination,
Geometric mean concentration (GMC) of IgG antibodies to 23 pneumococcal serotypes on 30 days after vaccination | 30 days
  Geometric mean concentration (GMC) of IgG antibodies to 23 pneumococcal serotypes on 30 days after vaccination
Incidence of adverse reactions/events within 30 minutes of vaccination | 30 min after vaccination
  Incidence of adverse reactions/events within 30 minutes of vaccination
Incidence of adverse reactions/events on days 0 to 7 after vaccination | 7 days
  Incidence of adverse reactions/events on days 0 to 7 after vaccination
Incidence of adverse reaction/event on days 0 to 30 after vaccination | 30 days
  Incidence of adverse reaction/event on days 0 to 30 after vaccination
Incidence of serious adverse events (SAE) within 6 months after vaccination | 6 months
  Incidence of serious adverse events (SAE) within 6 months after vaccination

SECONDARY OUTCOMES:
Geometric mean fold increase (GMFI) of IgG antibodies against 23 pneumococcal serotypes 30 days after vaccination | 30 days
  Geometric mean fold increase (GMFI) of IgG antibodies against 23 pneumococcal serotypes 30 days after vaccination
GMC of 23 pneumococcal serotype IgG antibodies in the 3rd and 6th year after vaccination | 3, 6 years after vaccination
  GMC of 23 pneumococcal serotype IgG antibodies in the 3rd and 6th year after vaccination

OTHER OUTCOMES:
The proportion of subjects with ≥0.35ug/mL IgG antibodies to 23 pneumococcal serotypes 30 days after vaccination, | 30 days
  The proportion of subjects with ≥0.35ug/mL IgG antibodies to 23 pneumococcal serotypes 30 days after vaccination,

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Center For Disease Control and Prevention, Chengdu, Sichuan, China